CLINICAL TRIAL: NCT01291498
Title: High Intensity Focused Ultrasound (HIFU) for Parathyroid Adenoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The manufacturer is not currently supporting research in this indication.
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-PT-2010-01
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2014-07

CONDITIONS: Parathyroid Adenomas
Keywords: Primary Parathyroid Adenomas
MeSH Terms: conditions — Parathyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU Treatment (Other): High Intensity Focused Ultrasound. This is not a comparative study
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — One or two HIFU sessions
  Other Names: TH-One HIFU device

SUMMARY:
This study aims to determine whether HIFU treatment is a safe and effective alternative to an operation to remove all or part of the affected gland. The objective is to achieve biochemical cure (assessed by normal calcium level in the blood at six weeks, six months and one year after therapy) without affecting the patient's voice or ability to swallow.

DETAILED DESCRIPTION:
Primary hyperparathyroidism is a common endocrine condition in which one or more of the four parathyroid glands in the neck releases too much parathyroid hormone (PTH). this leads to excess calcium in the blood and if untreated it can cause osteoporosis, kidney stone formation, deterioration of kidney function and disturbance in heart rhythm. Surgery to remove all or part of the affected gland(s) is expected to cure 95% of such patients. In current practice all such patients undergo localisation techniques using sestamibi scanning and neck ultrasonography to demonstrate the position of the enlarged/overactive parathyroid gland. These radiological tests are positive in some two thirds of patients, who can be operated through a minimally invasive procedure focused on the exact localisation pinpointed by the scans.

This study uses a procedure that does not require a surgical incision. Precise imaging of the parathyroid glands allows the exact position of the tumour to be found from outside the body. A High Intensity Focused Ultrasound beam produces heat, but only in a small specific area. Exact positioning of the ultrasound beam targets the tumour cells and kills them without harming the surrounding healthy tissues.

ELIGIBILITY:
Inclusion Criteria:

* Primary Hyperparathyroidism (PHPT)
* Moderate/severe hypercalcaemia (Ca>2.8mmol/L)
* Positive sestamibi scan demonstrating a cervical parathyroid adenoma
* Adenoma visible on ultrasound scan

Exclusion Criteria:

* Large adenoma (>15mm)
* Deep adenoma (>20mm from skin surface
* Familial disease (eg members of MEN-1 families)
* Inability to complete questionnaires in English without making mistakes or needing help with translation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radu Mihai, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient entered the study. Screening and informed consent was conducted on 19 April 2011 and treatment was conducted at the Churchill Hospital on 31 May 2011
Pre-assignment Details: The company manufacturing the device reviewed patient's images before confirming eligibility for treatment.
Groups:
- HIFU Treatment: This is a single arm study, all subjects are planned to receive HIFU treatment
Period: Overall Study
Arm/Group | HIFU Treatment
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- HIFU Treatment: This is a single arm study, all subjects are planned to received HIFU treatment
Arm/Group | HIFU Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (NA) — Only one subject entered the study
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Eucalcaemia
Description: Calcium in the blood is measured from venepuncture
Time Frame: 12 months post-treatment
Population: The primary endpoint was not analysed because only one subject was entered and this subject was withdrawn from the study before 12 months after treatment.
Arm/Group | HIFU Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Eucalcaemia
Description: Ca in plasma
Time Frame: Six weeks post-treatment.Six month data were also intended to be reported, however, six month data were not analyzed because only one subject was entered and this subject was withdrawn from the study before six months after treatment.
Population: Six month data were also intended to be reported, however, six month data were not analyzed because only one subject was entered and this subject was withdrawn from the study before six months after treatment.
Measure: Number; unit: mmol/L
Groups:
- HIFU Treatment: Ablation of the parathyroid gland by HIFU Treatment
Arm/Group | HIFU Treatment
Number analyzed (Participants) | 1
mmol/L | 1

3. Secondary Outcome: Voice Morbidity
Description: Voice Handicap Index. 30 questions rated on a five point scale from 'never' to 'always' and an overall score from 1 'normal' to 10 'severely impaired'
Time Frame: Up to one year post-treatment
Measure: Number; unit: units on a scale
Groups:
- HIFU Treatment: Allsubjects are planned to have HIFU Treatment
Arm/Group | HIFU Treatment
Number analyzed (Participants) | 1
units on a scale | 1

ADVERSE EVENTS:
Arm/Group | HIFU Treatment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes